CLINICAL TRIAL: NCT03310879
Title: A Phase II Study of the CDK4/6 Inhibitor Abemaciclib in Patients With Solid Tumors Harboring Genetic Alterations in Genes Encoding D-Type Cyclins or Amplification of CDK4 or CDK6
Brief Title: Study of the CDK4/6 Inhibitor Abemaciclib in Solid Tumors Harboring Genetic Alterations in Genes Encoding D-Type Cyclins or Amplification of CDK4 or CDK6
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Geoffrey Shapiro, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-343
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants with CCND1, CCND2, or CCND3 (Experimental): * Abemaciclib will be administered orally on a daily basis
  * Dosage will be determine by the PI
  Interventions: Drug: Abemaciclib
- Participants with CDK4 or CDK6 (Experimental): * Abemaciclib will be administered orally on a daily basis
  * Dosage will be determine by the PI
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib is a cyclin-dependent kinase (CDK) inhibitor. CDK inhibitors work to stop cell growth.

SUMMARY:
This research study is studying a targeted therapy as a possible treatment for cancer abnormality in one of the following genes: CCND1, CCND2, CCND3, CDK4, or CDK6.

The drug involved in this study is:

-Abemaciclib

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Abemaciclib as a treatment for any disease.

To participate in this study, the participant must have an abnormality in one of the following genes: CCND1, CCND2, CCND3, CDK4, or CDK6. Abnormalities in these genes may cause the cancer to grow more rapidly. CDK4 and CDK6 are proteins that are involved with the cell growth process. D-type cyclins (CCND1, CCND2, and CCND3) are proteins that help control the activity of CDK4 and CDK6.

Abemaciclib is being studied as a treatment for people with advanced cancer. Abemaciclib is a cyclin-dependent kinase (CDK) inhibitor. CDK inhibitors work to stop cell growth. In this research study, the investigators are hoping to learn whether Abemaciclib can be used to slow or stop the growth of cancers with specific genetic abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically or cytologically confirmed advanced solid tumor of a non-breast origin, for which standard therapy proven to provide clinical benefit does not exist or is no longer effective.
* For enrollment to Arm 1: Participants must have a confirmed CCND1, 2, or 3 high-level amplification, CCND1 mutation, or a CCND1 splice variant expected to lead to nuclear retention of cyclin D1 protein, via DFCI/BWH OncoPanel or any CLIA-certified method.
* For enrollment to Arm 2: Participants must have a confirmed CDK4 or CDK6 high-level amplification, identified via DFCI/BWH OncoPanel or any CLIA-certified method.
* Participants must have evaluable or measurable disease.
* Age ≥ 18 years.
* ECOG performance status of 0-1 (see APPENDIX A).
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional (ULN) -OR-
  * AST(SGOT)/ALT(SGPT) ≤ 5 × institutional (ULN) if liver metastases are present
  * Serum Creatinine ≤ 1.5 × institutional ULN -OR-
  * Creatinine clearance ≥ 60 mL/min (Cockroft-Gault Equation)
* The effects of abemaciclib on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 3 months after completion of abemaciclib administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. A negative serum pregnancy test is required for women of childbearing potential prior to study entry.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* Participants who have had chemotherapy, biologic therapy, investigational agents, radiotherapy, or major surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Participants who have had oral targeted therapy or oral tyrosine kinase inhibitors (TKIs) within 5 half-lives prior to entering the study.
* Participants who have received prior treatment with a CDK4/6 inhibitor.
* Participants must have recovered to eligibility levels from prior toxicity or adverse events as a result of previous treatment prior to entering the study.
* Participants who are receiving any other investigational agents.
* Participants with hematologic lymphoma.
* Participants with symptomatic CNS metastases who are neurologically unstable and/or require radiation therapy are excluded.

  * Participants with brain metastases that do not meet the above criteria in the opinion of the treating investigator are allowed.
  * Symptomatic disease is allowed as long as symptoms are controlled and stable.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to abemaciclib.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because abemaciclib is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with abemaciclib, breastfeeding should be discontinued if the mother is treated with abemaciclib. A negative serum pregnancy test is required for women of childbearing potential prior to study entry.
* Participants with known HIV-positive status are ineligible because these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Participants with known active Hepatitis B or Hepatitis C.
* Participants receiving an enzyme-inducing antiepileptic drug (EIAED) who cannot be transferred to a non-EIAED (e.g., levetiracetam, lacosamide, lamotrigine, etc.) prior to the initiation of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2017-11-21 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Rate | 4 months
  proportion of patients who are alive and progression-free at 4 months on both arms.

SECONDARY OUTCOMES:
Overall Response Rate | 2 years
  objective response rate by RECIST 1.1 for patients enrolled to both arms.
Toxicity | 2 years
  Adverse event data in all participants by CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No